CLINICAL TRIAL: NCT05296538
Title: The Mental Imagery for Suicidality in Students Trial (MISST): A Feasibility Study.
Brief Title: The Mental Imagery for Suicidality in Students Trial (MISST)
Acronym: MISST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Greater Manchester Mental Health NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Peter Taylor, Senior Clinical Lecturer, Greater Manchester Mental Health NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: x557s IRAS 305348
Record Dates: First submitted 2022-02-11; First posted 2022-03-25 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation | interventions — Risk Assessment

STUDY DESIGN:
Intervention Model Description: The MISST study is a two-armed feasibility randomised controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Researchers conducting assessments will be masked to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broad-Minded Affective Coping Intervention + Risk assessment and signposting (Experimental): Participants will first receive one to two 50 minute sessions focused on risk assessment and management, including signposting to further support. They will then be offered six sessions of the Broad-Minded Affective Coping (BMAC) Intervention. Sessions will take place weekly where possible and the intervention window will be eight weeks. A booster session will be offered in the 8 weeks following the end of therapy.
  Interventions: Other: Broad-Minded Affective Coping Intervention; Other: Risk Assessment and Signposting
- Risk assessment and signposting + Treatment As Usual (Other): Participants will first receive one to two 50 minute sessions focused on risk assessment and management, including signposting to further support. In addition they will be able to access usual care from their University counselling service or other health services.
  Interventions: Other: Risk Assessment and Signposting

INTERVENTIONS:
Other: Broad-Minded Affective Coping Intervention — The Broad-Minded Affective Coping (BMAC) is a six session intervention that uses mental imagery and rehearsal of memories of past positive experiences to generate positive emotions in the moment. A further follow-up session is provided in the eight weeks following the end of treatment.
  Arms: Broad-Minded Affective Coping Intervention + Risk assessment and signposting
Other: Risk Assessment and Signposting — A therapist will meet with participants over two 50 minute sessions to conduct a comprehensive risk assessment, and develop a collaborative plan with the participant around managing any risk, including identification of sources of support and signposting.

SUMMARY:
In the UK, suicide is the leading cause of death in young people and have increased in recent years. Areas in the North of England appear particularly at risk. University students represent one vulnerable group. 42% of students contemplate suicide in any one-year period. Suicidal thinking is an important indicator of distress and clinical need, which predicts subsequent suicidal experiences and worse mental health. It is therefore an important target for clinical treatment and early intervention. However, evidenced based interventions for targeting suicidal thinking in students are lacking.

This project will evaluate the feasibility of a novel psychological intervention, called the Broad Minded Affective Coping (BMAC) intervention. The BMAC aims to increase peoples' access to positive thoughts and emotions to help them to break out of cycles of negative mood and suicidal thinking. It is targeted, protocolised, and deliverable by a range of professional groups. Our existing co-development work with young people has suggested that it is acceptable and helpful to University students. This randomised controlled feasibility trial of the BMAC intervention for suicidal thinking in university students. Participants will be randomised to either a risk assessment and signposting plus the BMAC (n = 33), or risk assessment and signposting alone (n = 33). The study will assess outcomes at baseline and after eight weeks, 16 weeks, and 24 weeks. The study will explore the safety, feasibility and acceptability of delivering the intervention and trial procedures. Embedded qualitative interviews with staff and participants, and field notes, will help us to understand the potential factors affecting acceptability and delivery of the BMAC intervention and conduct of the trial, and the proposed underlying mechanisms of change. The project will be a crucial step in evaluating the BMAC for suicidal students, paving the way for a larger trial of clinical effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* Accessing full or part time education through a Higher Education Institution (HEI).
* Suicidal ideation and/or behaviours in the past three months

Exclusion Criteria:

* Active/historical full threshold first episode psychosis or bipolar disorder
* Known moderate to severe learning disability (IQ:<70).
* Organic cerebral disease/injury affecting receptive and expressive language comprehension.
* Non-English speaking to the degree that the participant is unable to answer questions and give written informed consent.
* Imminent and immediate risk to self or others, operationalised as the presence of active intent or planning to harm oneself or others in the near future (e.g. next month).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Recruitment Rates | 2 years
  Ability to randomise 66 participants in an 11-month recruitment window. Traffic light targets for the percentage of the target sample recruited is as follows: Green: ≥80%. Amber 60-<80%. Red <60%.
Adherence to treatment | 24 weeks
  Percentage of participants receiving the minimum dose of BMAC therapy (≥2 sessions) within eight-week treatment window. Traffic light targets for the percentage of the target sample receiving the minimum dose is as follows: Green: ≥80%. Amber: 60-<80%. Red: <60%.
Suitability of proposed primary outcome | Through study completion, an average of 24 weeks
  Informed by qualitative workstream plus percentage of participants completing the Beck Scale for Suicidal ideation y(BSS) at all timepoints. Targets for the proportion of participants completing the BSS is as follows: Green: ≥80%. Amber: 60-<80%. Red: <60%.
Occurrence of Adverse Reactions | Through study completion, an average of 24 weeks
  Monitoring and review of research related serious adverse events (SAEs). The Trial Steering Committee (TSC) will oversee SAEs across treatment arms.

SECONDARY OUTCOMES:
Beck Scale of Suicidal Ideation (BSS) | Baseline, 8-weeks, 16-weeks, 24-weeks
  This is a 21-item questionnaire measuring suicidal thinking over the past week. Items are scored on a scale from 0 to 2, with total scores ranging from 0 to 38, higher scores indicating greater suicidal ideation.
Beck Hopelessness Scale (BHS) | Baseline, 8-weeks, 16-weeks, 24-weeks
  This is a 20-item questionnaire measuring feelings of hopelessness over the past week. Items are scored on a scale from 0 to 1 (true or false), with total scores ranging from 0 to 20, higher scores indicating greater hopelessness.
Defeat and Entrapment Scale short-form (DES - short) | Baseline, 8-weeks, 16-weeks, 24-weeks
  This is an 8-item questionnaire measuring feelings of defeat and entrapment. Items are scored on a scale from 0 to 4, with total scores ranging from 0 to 32, higher scores indicating greater perceived defeat and entrapment.
Generalised Anxiety Disorder Assessment (GAD-7) | Baseline, 8-weeks, 16-weeks, 24-weeks
  This is a 7-item questionnaire measuring anxiety symptoms over the preceding two weeks. Items are scored on a scale from 0 to 3, with total scores ranging from 0 to 21, higher scores indicating greater anxiety.
Positive and Negative Affect Schedule (PANAS) | Baseline, 8-weeks, 16-weeks, 24-weeks
  This is a 20-item questionnaire measuring positive and negative affective states. Items are scored on a scale from 0 to 5, with total scores ranging from 0 to 50 for the negative affect and positive affect subscales, where higher scores indicating experience of greater positive and negative affect, respectively.
Perceived Control of Internal States Scale (PCISS) | Baseline, 8-weeks, 16-weeks, 24-weeks
  This is an 18-item questionnaire measuring perceived control of internal states (e.g. emotions and cognitions). Items are scored on a scale from 1 to 5, with total scores ranging from 18 to 90, where higher scores indicating greater perceived control.
Patient Health Questionnaire (PHQ9) | Baseline, 8-weeks, 16-weeks, 24-weeks
  This is a 9-item questionnaire measuring depressive symptoms over the preceding two weeks. Items are scored on a scale from 0 to 3, with total scores ranging from 0 to 27, where higher scores indicating greater depression.
Perceived Stress Scale (PSS) | Baseline, 8-weeks, 16-weeks, 24-weeks
  This is a 10-item questionnaire measuring stress over the preceding month. Items are scored on a scale from 0 to 4, with total scores ranging from 0 to 40, where higher scores indicating greater stress.
The Self-Injurious Thoughts and Behaviours Interview (SITBI) + Linehan Suicide Attempt-Self-Injury Interview (SASII) | Baseline, 8-weeks, 16-weeks, 24-weeks
  The SITBI is a structured interview designed to assess self-injurious and suicidal thoughts and behaviours. The sections relating to suicide attempt and non-suicidal self-injury will be used. In these sections the frequency of suicidal and self-injurious behaviour over the preceding year, month, and week is assessed. These data on occurrence of suicidal and self-injurious behaviour will be used as a secondary outcome in the trial. Items adapted from the SASII regarding the frequency of self-harm occurring over one's life and since the last assessment, will also be used to supplement the SASII in assessing suicidal and self-injurious behaviour. Frequency of suicidal or self-harm behaviour since the previous assessment point will be recorded at each follow-up assessment using these measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Greater Manchester Mental Health NHS Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palmier-Claus J, Duxbury P, Pratt D, Parker S, Sutton C, Lobban F, Moorhouse J, Kerry E, Russell C, Nyakutsikwa B, Drake R, Eccles S, Randles N, Patel R, Kelly J, Tattersall R, Taylor PJ. A mental imagery intervention targeting suicidal ideation in university students: An assessor-blind, randomised controlled feasibility trial. Behav Res Ther. 2025 Aug;191:104780. doi: 10.1016/j.brat.2025.104780. Epub 2025 May 20. PMID 40411963
- [Derived] Taylor PJ, Duxbury P, Moorhouse J, Russell C, Pratt D, Parker S, Sutton C, Lobban F, Drake R, Eccles S, Ryder D, Patel R, Kimber E, Kerry E, Randles N, Kelly J, Palmier-Claus J. The Mental Imagery for Suicidality in Students Trial (MISST): study protocol for a feasibility randomised controlled trial of broad-minded affective coping (BMAC) plus risk assessment and signposting versus risk assessment and signposting alone. Pilot Feasibility Stud. 2023 Mar 17;9(1):43. doi: 10.1186/s40814-023-01273-7. PMID 36932430